CLINICAL TRIAL: NCT06348017
Title: Frequency of Neuropathic Pain and Central Sensitization in Patients With Plantar Fasciitis
Brief Title: Frequency of Neuropathic Pain in Patients With Plantar Fasciitis
Status: Completed | Type: Observational
Sponsor: Yozgat City Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Yozgat City Hospital
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Chronic Plantar Fasciitis; Control Group
Keywords: Plantar fasciitis; Neuropathic pain; Central sensitization; Pain-DETECT; Central Sensitization Scale; Foot Function Index
MeSH Terms: conditions — Fasciitis, Plantar; Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Design This prospective cross-sectional study was undertaken between November 2023 and March 2024. Written and verbal informed consent was obtained from all patients. The study protocol was approved by University Human Research Ethics Committee (AEŞH-EK 1-2023-612).

Patients While 106 patients who applied to the City Hospital Physical Medicine and Rehabilitation outpatient clinic with heel pain that had been present for at least six months, received foot radiography and were diagnosed with PF were included in the study as a patient group; 100 patients who did not have foot pain and had musculoskeletal pain for at least 6 months were included in the study as a control group, between November 2023 and March 2024. All the participants were aged 18 to 65 years. Patients with a history of diabetes, hypothyroidism and CKD, a history of malignancy, with vasculitis, neurological diseases that may cause neuropathic pain, lumbar discopathy, those with a previous history of fracture or surgery in the heel area, received injections or ESWT treatment due to heel pain in the last 3 months, rheumatic diseases that may affect pain such as rheumatoid arthritis, ankylosing spondylitis, fibromyalgia, and severe circulatory disorders on the side with pain, were excluded from the study. The study was commenced after obtaining the approval of the local ethics committee and informed consent of the participants.

All patients' personal information (age, gender, occupation, education information), general health information (smoking and alcohol use information, known chronic disease history, body mass index), severity of heel pain and when it started were recorded. While the Foot Function Index (FFI) scale, which evaluates the functionality of the foot, was applied to the patient group; the Visual Analog Scale (VAS), which evaluates pain intensity, the Pain-DETECT scale, which evaluates neuropathic pain, and the Central Sensitization Scale (CSI), which evaluates central sensitization, were applied to the patient and control groups. The details of the implementation of the instruments are as follows:

DETAILED DESCRIPTION:
Visual Analog Scale (VAS) for the Evaluation of Pain and Fatigue For this evaluation, the patient is asked to mark his/her severity of pain and fatigue on a horizontal 10-cm line with number 0 on one end representing "no pain or no fatigue" and number 10 on the other end indicating "very severe pain or very severe fatigue".

Foot Function Index (FFI): Sub-parameters of FFI; pain, disability and activity limitation and is a scale consisting of a total of 23 items. The pain subscale includes nine items and measures the severity of foot pain in different situations. The disability subscale includes 9 items and evaluates the severity of the person's difficulty in performing functional activities due to foot problems. The activity limitation subscale includes 5 items and measures the person's activity limitations due to foot problems. People answer the questions with the Visual Analogue Scale (VAS), taking into account their foot conditions a week ago. A higher score indicates more pain, disability, and activity limitation. Turkish validity and reliability study was conducted by Yalıman et al. in 2014.

Pain-DETECT: The survey consists of 9 questions, with a score range of 1-38. Scores of 12 and below are considered as 'NA component is unlikely', scores between 13-18 are considered as 'NA component is uncertain', and scores of 19 and above are considered as 'NA component is possible'. Turkish validity and reliability study was conducted by Alkan et al in 2013.

Central Sensitization Scale (CSI): The survey consists of 25 questions. Each question is scored between 0 and 4 (0=never, 4=always). A score of forty and above 31 indicates the presence of CS with 81% sensitivity and 75% specificity. SS severity is defined as 0-29 subclinical, 30-39 mild, 40-49 moderate, 50-59 severe, 60 and above very severe. Turkish validity and reliability study was conducted by Keleş et al in 2021.

ELIGIBILITY:
Inclusion Criteria:

* • Applied to the City Hospital Physical Medicine and Rehabilitation outpatient clinic with heel pain that had been present for at least six months

  * received foot radiography and were diagnosed with PF
  * aged 18 to 65 years as a patient group;
  * musculoskeletal pain for at least 6 months
  * who did not have foot pain
  * aged 18 to 65 years as a control group

Exclusion Criteria:

* A history of diabetes, hypothyroidism and congestive heart failure
* A history of malignancy
* Vasculitis
* Neurological diseases that may cause neuropathic pain,
* Lumbar discopathy
* A previous history of fracture or surgery in the heel area
* Received injections or ESWT treatment due to heel pain in the last 3 months
* Rheumatic diseases that may affect pain such as rheumatoid arthritis, ankylosing spondylitis, fibromyalgia
* Severe circulatory disorders on the side with pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who applied to the City Hospital Physical Medicine and Rehabilitation outpatient clinic with heel pain that had been present for at least six months, received foot radiography and were diagnosed with PF Patients who did not have foot pain and had musculoskeletal pain for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Pain-DETECT | One Time
  The survey consists of 9 questions, with a score range of 1-38. Scores of 12 and below are considered as 'NA component is unlikely', scores between 13-18 are considered as 'NA component is uncertain', and scores of 19 and above are considered as 'NA component is possible'. Turkish validity and reliability study was conducted by Alkan et al in 2013
Foot Function Index | One Time
  Sub-parameters of FFI; pain, disability and activity limitation and is a scale consisting of a total of 23 items. The pain subscale includes nine items and measures the severity of foot pain in different situations. The disability subscale includes 9 items and evaluates the severity of the person's difficulty in performing functional activities due to foot problems. The activity limitation subscale includes 5 items and measures the person's activity limitations due to foot problems. People answer the questions with the Visual Analogue Scale (VAS), taking into account their foot conditions a week ago. A higher score indicates more pain, disability, and activity limitation. Turkish validity and reliability study was conducted by Yalıman et al. in 2014
Central Sensitization Scale | One Time
  The survey consists of 25 questions. Each question is scored between 0 and 4 (0=never, 4=always). A score of forty and above 31 indicates the presence of central sensitization with 81% sensitivity and 75% specificity. SS severity is defined as 0-29 subclinical, 30-39 mild, 40-49 moderate, 50-59 severe, 60 and above very severe (12). Turkish validity and reliability study was conducted by Keleş et al in 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Yozgat City Hospital, Yozgat, Turkey (Türkiye)